CLINICAL TRIAL: NCT02905474
Title: Harnessing Mobile Health Technology to Personalize the Care of Chronic Kidney Disease Patients: Medication Domain Randomized Controlled Trial
Brief Title: Mobile Health Technology for Chronic Kidney Disease Patients: Medication Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UHN-16-5002-BE
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Renal Insufficiency, Chronic; Hypertension; Medication Reconciliation; Mobile Applications
Keywords: chronic kidney disease, mobile applications, mHealth, medication reconciliation, self-management
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- eKidneyCare (Experimental): The eKidneyCare mobile app has an active interface with the renal clinic pharmacy system to allow for updated medication profiles to be sent directly to the patient's smartphone for the renal clinic pharmacy information system.
  Interventions: Other: Usual Care; Device: Integrated mobile medication app
- My MedRec (Commercial App) (Active Comparator): My MedRec is a commercially available mobile app which allows a user to have a personal health record along with keeping track of their medications. The My MedRec mobile app allows users to track blood pressure and medication information through manual data entry with the app. It is a stand alone mobile app which stores specified medical information on the native smartphone device and does not connect to any other servers or databases.
  Interventions: Other: Usual Care; Device: Commercially available mobile medication app

INTERVENTIONS:
Other: Usual Care — Usual standard CKD care involves an outpatient clinic visit every 3 to 4 months (at minimum every 6 months) for a clinical assessment by their renal clinical care team.
Device: Integrated mobile medication app — Use of mobile app to maintain, manage medication list on a smartphone device that allows for bidirectional transfer of medication information
  Arms: eKidneyCare
Device: Commercially available mobile medication app — Use of mobile app to manually record and maintain medication records with no integration to databases.
  Arms: My MedRec (Commercial App)

SUMMARY:
Patients with complex, long-lasting conditions such as chronic kidney disease (CKD) often take multiple medications and frequently have serious medication problems, arising from poor communication between doctors and patients. Prescription errors or misunderstandings can cause harm and lead to emergency room visits or even hospitalizations. To address these issues, medication reconciliation is now used by hospitals as a way to confirm the medication list of patients on admission to and discharge from hospital. However, a similar process does not exist outside the hospital setting. In recent years patients have become more proactive in undertaking activities with a direct bearing on their health. Such activities may include maintaining an accurate list of their medications. The rapid growth of the digital health arena has led to the development of a large number of commercially available mobile medication management apps for patients. These digital tools are 'stand-alone' products that are not integrated with the patients' pharmacy or health record system. They rely on patients to enter the list of their medications and update it as necessary. Moreover, few have a function to communicate medication changes or problems with their healthcare providers. Recently, an integrated smartphone, eKidneyCare, app system was developed with a medication management feature to help patients maintain an accurate mobile medication list. Patients' current medication information in the pharmacy database is uploaded onto their by a pharmacist and changes are tracked regularly through a bi-directional communication system. Updates to the medication list occur seamlessly by the pharmacist, and patients and their physicians are notified about any medication errors or serious adverse events. This study will determine whether our eKidneyCare app with its medication management feature will decrease medication errors and improve patient safety compared to the more traditional way of managing medications.

DETAILED DESCRIPTION:
Background: Patients who have complicated conditions such as chronic kidney disease (CKD) are at high risk for problems related to their medications. Often these problems occur because doctors and patients do not communicate the right type of medication information to each other. This causes many prescribing errors and can lead to patient harm, emergency visits, or hospitalizations. To address this communication problem, hospitals now use a process called "medication reconciliation" to confirm the medications patients are taking when they enter and leave the hospital. However, the way that medication reconciliation is currently being done, patients are not actively engaged or given tools to effectively communicate the medications they are taking, changes that have been made, and what they are having trouble with. Directly engaging patients in this process might help solve this problem, and mobile technologies on smartphones may be a solution. Our study team has developed a mobile application (app) called eKidneyCare, which has a specific medication component to help patients communicate their medication information to all their doctors. This app can feed medication information from the clinic's medical record to the patient's smartphone, and any changes made to the medication list can be entered by the patient and sent back to the central server to notify their doctors.

Study Design: We propose to conduct an open-label randomized controlled trial to assess the medication related effectiveness and stakeholders' satisfaction of the eKidneyCare mobile app compared to commercially available mobile apps like My MedRec for 12 months. This study will be conducted in the renal clinics at University Health Network who oversee the clinical management of advanced stage 4 to 5 CKD patients and end stage renal disease. On average, patients of this clinic are aged 65 years or more and take 10-15 medications per day.

Objectives and Hypotheses Primary 1) To evaluate the effect of the eKidneyCare mobile app compared to a commercially available stand alone mobile app (My MedRec) on unintentional medication discrepancies in CKD patients. The use of the eKidneyCare app will have a greater reduction medication discrepancy rates by enhancing patient self-care through bidirectional communication of information.

Secondary

1. To determine the effect of the eKidneyCare mobile app compared to commercially available stand along mobile app (My MedRec) on CKD-specific clinical outcomes. Patients actively engaged in medication management will translate to improved clinical parameters such as better blood pressure control.
2. To evaluate the direct costs and quality of life (QOL) associated with incorporating the eKidneyCare mobile app compared to commercially available stand along mobile app (My MedRec). Reduction in the unintentional medication discrepancy rate will offset the cost of using the medication self-care app and will improve patients' quality of life.
3. To assess stakeholders' satisfaction in using the mobile app to manage CKD. Medication self-care app will increase satisfaction among patients.

This study will evaluated if this app will decrease errors related to medications. It is hypothesized that if patients use this app to report their medications to their doctors, fewer errors will occur, which should eventually lead to reduced patient harm and healthcare use.

ELIGIBILITY:
Inclusion Criteria:

* Incident or prevalent patients who are: ≥18 years of age
* English-speaking
* Able and willing to provide informed consent

Exclusion Criteria:

* CKD stages 1 to 3a (estimated glomerular filtration rate of ≥ 45 ml/min)
* likely to receive a kidney transplant within 3 months of enrollment into the trial
* living in a long-term care or rehabilitation institution, likely to have their care transferred to another facility outside participating clinic areas during the course of the study
* taking less than 2 prescription medications
* planning to travel or live consecutively out of the province of Ontario for more than one month
* participating in another intervention trial,
* cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2016-05; Primary Completion 2017-09-26 (Actual); Study Completion 2017-09-26 (Actual)

PRIMARY OUTCOMES:
Medication Discrepancy | One year (12 months)
  The change in unintentional medication discrepancy rate from baseline to the last (12 months) visit.

SECONDARY OUTCOMES:
Clinic Blood Pressure | 6, 12 months
  Mean change in systolic and diastolic BP measured by clinic BP Tru automated machine
Ambulatory Blood Pressure | 12 months
  Mean change in systolic and diastolic BP measured by average 7 day home ambulatory BP readings
CKD specific laboratory values (hemoglobin) | 12 months
  Proportion of patients in target hemoglobin, defined as hemoglobin of 100 to 120 g/L
CKD specific laboratory values (potassium) | 12 months
  Proportion of patients in target potassium ; defined as potassium of 3.2 to 5.0 mmol/L
CKD specific laboratory values (phosphate) | 12 months
  Proportion of patients in target phosphate; defined as phosphate range of less than 1.5 mmol/L.
Medication Discrepancy Proportion of Patients | 12 months
  Proportion of patients more than 1 unintentional discrepancy
Satisfaction | 12 months
  Key feedback on usability, experience and perceived strengths and weakness of mobile app
Quality of Life | 12 months
  Change in health utility scores as captured in the EQ-5D questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie W Ong, BScPHM, MSc, Principal Investigator — UHN; Alexander G Logan, MD, FRCP(C), Principal Investigator — Samuel Lunenfeld Research Institute, Mount Sinai Hospital
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ong SW, Jassal SV, Porter EC, Min KK, Uddin A, Cafazzo JA, Rac VE, Tomlinson G, Logan AG. Digital Applications Targeting Medication Safety in Ambulatory High-Risk CKD Patients: Randomized Controlled Clinical Trial. Clin J Am Soc Nephrol. 2021 Apr 7;16(4):532-542. doi: 10.2215/CJN.15020920. Epub 2021 Mar 18. PMID 33737321